CLINICAL TRIAL: NCT04803799
Title: Effects of an Exergame Focused on Cognitive-motor Interference on the Cognitive and Motor Capacities of Older Adults
Acronym: INCOME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 87RI20_0047 (INCOME)
Record Dates: First submitted 2021-03-08; First posted 2021-03-18 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2022-03

CONDITIONS: Ageing
Keywords: Cognitive, motor, abilities, exergame

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental Arm (Experimental): Training programme using Exergame as a support over a 12 week period
  Interventions: Other: Training Programme

INTERVENTIONS:
Other: Training Programme — Cognitive-motor dual task exercises corresponding to associations between different motor tasks and different cognitive tasks.

SUMMARY:
Ageing is accompanied by a high risk of developing physical or cognitive impairments, as well as a decrease in abilities to perform two tasks simultaneously, contributing to loss of autonomy.

Interventions based on the performance of cognitive-motor dual tasks show positive effects on cognitive, physical and emotional development on dual-tasking capabilities. Exergames, interactive serious games combining physical activity and technology, are a certain type of cognitive-motor dual task training. These exergames appear to be cognitively effective, discussed on a physical level, not studied on dual task functions. It is likely that a dual task cognitive-motor with the support of a exercise leads to the same benefits as training without the need for special support.

In addition, the exergames benefit from specific features such as a good immersion and a playful aspect that increase the participant's adhesion. Moreover, the level of security of this type of programme has been little studied. It is likely that cognitive-motor dual tasks training supported by an exercise programme leads to few undesirable events and good adherence.

Many of the recommendations specific needs gaming state that it is important to develop systems that respond to the needs specific to the population concerned in order to be effective. Within the laboratory HAVAE has been developed a tool, the "virtual carpet":

association between a video-projected scene and a monitoring system of position of the participants. This system makes it possible to use as a grid of play the cartography and iconography of the City of Limoges. The investigators suppose that this emphasis on local heritage will encourage the participants leaving their homes, thereby increasing their level of physical activity and their quality of life.

ELIGIBILITY:
Inclusion Criteria:

A person over 75 years of age who :

* resides in one of the two Municipal Autonomy Residences (RAM) of the City of Limoges (Durkheim or Casseaux), or a member of a senior club of the communal social action centre
* has normal or corrected vision and hearing

Exclusion Criteria:

Person presenting :

* psychiatric disorders or neurological pathologies (cardiovascular accidents, Parkinson's disease, Alzheimer's, dementia) diagnosed
* taking medication that affects walking or balance
* a need for technical assistance (double cane-crutch, walker)
* an inability to carry out the proposed training programme
* person unable to understand the Protocol

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Postural control under dual-task condition change | Week 3, Week 17
  assessed by posturography (mm/s)

SECONDARY OUTCOMES:
Mental inhibition under dual-task condition change | Week 3, Week 17, Week 31
  assessed by Stroop test time (s)
Mental inhibition under dual-task condition change | Week 3, Week 17, Week 31
  assessed by Stroop test errors (n)
Mental inhibition change single-task condition | Week 3, Week 17, Week 31
  assessed by Stroop test time (s)
Mental inhibition change single-task condition | Week 3, Week 17, Week 31
  assessed by Stroop test errors (n)
Mental flexibility change | Week 3, Week 17, Week 31
  assessed by TMT time (s)
Mental flexibility change | Week 3, Week 17, Week 31
  assessed by Stroop test errors (n)
Working memory change | Week 3, Week 17, Week 31
  assessed by 2N-Back test errors (n)
Mobility change | Week 3, Week 17, Week 31
  assessed by TUG time (s)
Balance change | Week 3, Week 17, Week 31
  assessed by BBS score
Fear of falling | Week 3, Week 17, Week 31
  assessed by FES-I score
Postural control under single-task condition change | Week 3, Week 17, Week 31
  assessed by posturography (mm/s)
Reported physical activity level change | Week 3, Week 17, Week 31
  assessed by QAPPA score
Traqued physical activity level change | Week 3, Week 17, Week 31
  assessed by embeded Armband
City exploration change | Week 17, Week 31
  assessed by the city's points of interest visits
Quality of life change | Week 3, Week 17, Week 31
  assessed by EQ5D5L score
Safety features of the training programme | Week 17
  number, nature, severity and causes of the occurrence of adverse events during the intervention
Compliance | Week 17
  assessed by number of sessions carried out
Drop-out | Week 17
  assessed by the number of participants who do not complete the program
Motivation change | Week 3, Week 17, Week 31
  assessed by EMAPS score

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Résidence Autonomie CASSEAUX, Limoges
  - Résidence Autonomie DURKHEIM, Limoges

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gallou-Guyot M, Mandigout S, Marie R, Robin L, Daviet JC, Perrochon A. Feasibility and potential cognitive impact of a cognitive-motor dual-task training program using a custom exergame in older adults: A pilot study. Front Aging Neurosci. 2023 Feb 2;15:1046676. doi: 10.3389/fnagi.2023.1046676. eCollection 2023. PMID 36819724